CLINICAL TRIAL: NCT03801317
Title: The Effect of Bovine Colostrum/ Egg Supplementation in Young Malawian Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Project Peanut Butter (Other); Kamuzu University of Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 201808199
Record Dates: First submitted 2019-01-10; First posted 2019-01-11 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Stunting; Environmental Enteric Dysfunction
MeSH Terms: conditions — Growth Disorders | interventions — Eggs

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BC/ egg (Experimental): 4.3 grams egg powder + 5.7 grams bovine colostrum
  Interventions: Dietary Supplement: BC/ egg; Dietary Supplement: multiple micronutrient
- Control (Placebo Comparator): 15 grams corn-soya blend
  Interventions: Dietary Supplement: Control; Dietary Supplement: multiple micronutrient

INTERVENTIONS:
Dietary Supplement: BC/ egg — 4.3 egg powder + 5.7 g bovine colostrum
  Arms: BC/ egg
Dietary Supplement: Control — 15 grams corn-soya blend
  Arms: Control
Dietary Supplement: multiple micronutrient — multiple micronutrient sprinkle powder

SUMMARY:
The trial will consist of adding either a supplement of 4.3g egg powder + 5.7g bovine colostrum or a control flour along with a multiple micronutrient powder to the diets of healthy Malawian children 9 months of age. This supplement provides additional essential amino acids, choline and immunoactive colostrum. Children will be receive either the supplement or control for 12 weeks. Children will have regular follow-up where anthropometry is measured. At enrollment and after 12 weeks, stool will be collected and a urinary lactulose permeability test conducted. Children will be measured at enrollment and at weeks 2, 4, 8, 12, 20, 32 after enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Children at 9-10 months of age

Exclusion Criteria:

* Malnutrition
* congenital abnormalities
* chronic diseases such as heart disease, cerebral palsy, or HIV infection

Ages: 9 Months to 10 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 278 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Intestinal permeability | 12 weeks
  The lactulose permeability test involves drinking 20 mL of a sugar water solution and collecting urine for 4 hours thereafter
Linear growth | 12 weeks and 32 weeks
  Change in length expressed as anthropometric z-score from enrollment to end point

SECONDARY OUTCOMES:
Incidence of diarrhea | 12 weeks
  Caregiver report of number of days they child has diarrhea over the course of the study
Adverse effects of the bovine colostrum/ egg | 12 weeks
  Caregiver report of number of days they child has adverse effects over the course of the study
16S configuration of fecal microbiota | 12 weeks
  Looking at the 16S configuration in stool samples collected
Stunting | 12 and 32 weeks
  Categorization of length-for-age z-scores
Environmental enteric dysfunction | 12 weeks
  Categorization of lactulose permeability measurements

CONTACTS AND LOCATIONS:
Locations (1):
- Project Peanut Butter, Malawi, Blantyre, Malawi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Owino V, Ahmed T, Freemark M, Kelly P, Loy A, Manary M, Loechl C. Environmental Enteric Dysfunction and Growth Failure/Stunting in Global Child Health. Pediatrics. 2016 Dec;138(6):e20160641. doi: 10.1542/peds.2016-0641. Epub 2016 Nov 4. PMID 27940670
- [Background] Prendergast AJ, Humphrey JH. The stunting syndrome in developing countries. Paediatr Int Child Health. 2014 Nov;34(4):250-65. doi: 10.1179/2046905514Y.0000000158. Epub 2014 Oct 13. PMID 25310000
- [Background] McKay S, Gaudier E, Campbell DI, Prentice AM, Albers R. Environmental enteropathy: new targets for nutritional interventions. Int Health. 2010 Sep;2(3):172-80. doi: 10.1016/j.inhe.2010.07.006. PMID 24037697
- [Background] Ordiz MI, Stephenson K, Agapova S, Wylie KM, Maleta K, Martin J, Trehan I, Tarr PI, Manary MJ. Environmental Enteric Dysfunction and the Fecal Microbiota in Malawian Children. Am J Trop Med Hyg. 2017 Feb 8;96(2):473-476. doi: 10.4269/ajtmh.16-0617. Epub 2016 Dec 12. PMID 27956653
- [Background] Semba RD, Trehan I, Li X, Moaddel R, Ordiz MI, Maleta KM, Kraemer K, Shardell M, Ferrucci L, Manary M. Environmental Enteric Dysfunction is Associated with Carnitine Deficiency and Altered Fatty Acid Oxidation. EBioMedicine. 2017 Mar;17:57-66. doi: 10.1016/j.ebiom.2017.01.026. Epub 2017 Jan 18. PMID 28122695
- [Background] Semba RD, Gonzalez-Freire M, Moaddel R, Trehan I, Maleta KM, Khadeer M, Ordiz MI, Ferrucci L, Manary MJ. Environmental Enteric Dysfunction Is Associated With Altered Bile Acid Metabolism. J Pediatr Gastroenterol Nutr. 2017 Apr;64(4):536-540. doi: 10.1097/MPG.0000000000001313. PMID 27322559
- [Background] Semba RD, Shardell M, Sakr Ashour FA, Moaddel R, Trehan I, Maleta KM, Ordiz MI, Kraemer K, Khadeer MA, Ferrucci L, Manary MJ. Child Stunting is Associated with Low Circulating Essential Amino Acids. EBioMedicine. 2016 Apr;6:246-252. doi: 10.1016/j.ebiom.2016.02.030. Epub 2016 Feb 19. PMID 27211567
- [Background] Semba RD, Zhang P, Gonzalez-Freire M, Moaddel R, Trehan I, Maleta KM, Ordiz MI, Ferrucci L, Manary MJ. The association of serum choline with linear growth failure in young children from rural Malawi. Am J Clin Nutr. 2016 Jul;104(1):191-7. doi: 10.3945/ajcn.115.129684. Epub 2016 Jun 8. PMID 27281303
- [Background] Semba RD, Shardell M, Trehan I, Moaddel R, Maleta KM, Ordiz MI, Kraemer K, Khadeer M, Ferrucci L, Manary MJ. Metabolic alterations in children with environmental enteric dysfunction. Sci Rep. 2016 Jun 13;6:28009. doi: 10.1038/srep28009. PMID 27294788
- [Background] Semba RD, Trehan I, Gonzalez-Freire M, Kraemer K, Moaddel R, Ordiz MI, Ferrucci L, Manary MJ. Perspective: The Potential Role of Essential Amino Acids and the Mechanistic Target of Rapamycin Complex 1 (mTORC1) Pathway in the Pathogenesis of Child Stunting. Adv Nutr. 2016 Sep 15;7(5):853-65. doi: 10.3945/an.116.013276. Print 2016 Sep. PMID 27633102
- [Background] Iannotti LL, Lutter CK, Bunn DA, Stewart CP. Eggs: the uncracked potential for improving maternal and young child nutrition among the world's poor. Nutr Rev. 2014 Jun;72(6):355-68. doi: 10.1111/nure.12107. Epub 2014 May 7. PMID 24807641
- [Background] Saad K, Abo-Elela MGM, El-Baseer KAA, Ahmed AE, Ahmad FA, Tawfeek MSK, El-Houfey AA, Aboul Khair MD, Abdel-Salam AM, Abo-Elgheit A, Qubaisy H, Ali AM, Abdel-Mawgoud E. Effects of bovine colostrum on recurrent respiratory tract infections and diarrhea in children. Medicine (Baltimore). 2016 Sep;95(37):e4560. doi: 10.1097/MD.0000000000004560. PMID 27631207
- [Background] Halasa M, Maciejewska D, Baskiewicz-Halasa M, Machalinski B, Safranow K, Stachowska E. Oral Supplementation with Bovine Colostrum Decreases Intestinal Permeability and Stool Concentrations of Zonulin in Athletes. Nutrients. 2017 Apr 8;9(4):370. doi: 10.3390/nu9040370. PMID 28397754
- [Background] Savarino SJ, McKenzie R, Tribble DR, Porter CK, O'Dowd A, Cantrell JA, Sincock SA, Poole ST, DeNearing B, Woods CM, Kim H, Grahek SL, Brinkley C, Crabb JH, Bourgeois AL. Prophylactic Efficacy of Hyperimmune Bovine Colostral Antiadhesin Antibodies Against Enterotoxigenic Escherichia coli Diarrhea: A Randomized, Double-Blind, Placebo-Controlled, Phase 1 Trial. J Infect Dis. 2017 Jul 1;216(1):7-13. doi: 10.1093/infdis/jix144. PMID 28541500
- [Derived] Bierut T, Duckworth L, Grabowsky M, Ordiz MI, Laury ML, Callaghan-Gillespie M, Maleta K, Manary MJ. The effect of bovine colostrum/egg supplementation compared with corn/soy flour in young Malawian children: a randomized, controlled clinical trial. Am J Clin Nutr. 2021 Feb 2;113(2):420-427. doi: 10.1093/ajcn/nqaa325. PMID 33330913